CLINICAL TRIAL: NCT04457479
Title: APERIO® HYBRID Thrombectomy Device for Flow Restoration in Vessels of Patients Experiencing Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Acandis GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: HYBRID
Record Dates: First submitted 2019-12-10; First posted 2020-07-07 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, multicenter, single-arm, open-label, national Post-Market Clinical Follow-up study to collect comprehensive information on technical and clinical success and safety of the use of APERIO® Hybrid(17/21) Thrombectomy Device in clinical practice. APERIO® Hybrid(17/21) Thrombectomy Device will be used within its approved indication.

DETAILED DESCRIPTION:
German APERIO® Hybrid Post- Market Clinical Follow-up Study

APERIO® Hybrid PMCF Study- Thrombectomy device for flow restoration in vessels of patients experiencing acute ischemic stroke

Study Type: prospective, multicenter, single-armed, open-label

Participants: 8 participating centers in Germany

PI: Dr. Christian Mathys, Evangelisches Krankenhaus Oldenburg, Germany

Estimated Enrolment: 190 patients treated with APERIO® HYBRID(17/21) Thrombectomy Device as a result of an acute stroke

Follow up: 3 months

Estimated Final Assessment: Mid to End of 2023

ELIGIBILITY:
Inclusion Criteria:

- All patients treated with APERIO® HYBRID and/or APERIO® Hybrid(17/21) Thrombectomy Device as a result of an acute stroke.

Exclusion Criteria:

* Patient age < 18 years
* Pre stroke mRS ≥ 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with acute large vessel occlusion (stroke) treated with the APERIO® Hybrid(17/21) Thrombectomy Device.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Technical success | until 24 hours after intervention
  mTICI ≥ 2b after treatment with APERIO® HYBRID(17/21)
Good clinical outcome at 90 days | 90 days after intervention
  Modified Rankin Scale (mRS) < 3 (mRS 1= no symptoms/ good outcome; mRS 6= Patient died/ worse outcome)
Periprocural symptomatic intracranial hemorrhage (sICH): | until 24 hours after intervention
  ICH in postinterventional (<24 hours) CT associated with worsening of NIHSS by ≥ 4 points within 24 hours

SECONDARY OUTCOMES:
Cerebrovascular events until hospital discharge: | between 24 hours after intervention and discharge from hospital
  * Intracranial haemorrhage (symptomatic / asymptomatic)
  * Death
  * TIA in the region of the target vessel
  * Non-disabling ischemic stroke (MRS 0-2) in the region of the target vessel
  * Disabling ischemic stroke (MRS 3-6) in the region of the target vessel
  * TIA outside the region of the target vessel
  * Non-disabling ischemic stroke (MRS 0-2) outside the region of the target vessel
  * Disabling ischemic stroke (MRS 3-6) outside the region of the target vessel
Cerebrovascular events at 90 days | at 90 days
  * Intracranial haemorrhage (symptomatic / asymptomatic)
  * Death
  * TIA
  * Non-disabling ischemic stroke (MRS 0-2)
  * Disabling ischemic stroke (MRS 3-6)

CONTACTS AND LOCATIONS:
Locations (1):
- Evangelisches Krankenhaus Oldenburg, Oldenburg, Germany